CLINICAL TRIAL: NCT03648944
Title: Accelerated vs Non-Accelerated Rehabilitation After Anterior Cruciate Ligament Reconstruction: A Pilot Study
Acronym: AVON ACL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: North Bristol NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R&I 3181
Record Dates: First submitted 2015-01-29; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2014-10

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Rehabilitation Outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Accelerated Rehabilitation (Experimental): Participants in this arm will have fewer restrictions on their mobility post-operatively and will be permitted to return to more active sporting activities quicker.
  Interventions: Other: Accelerated Rehabillitation
- Non-Accelerated (Active Comparator): Participants in this arm will be fitted with a knee brace and be restricted in their weight bearing post-operatively. They will also be restricted from returning to active sporting activities too quickly.
  Interventions: Other: Non-Accelerated Rehabillitation

INTERVENTIONS:
Other: Accelerated Rehabillitation
  Arms: Accelerated Rehabilitation
Other: Non-Accelerated Rehabillitation
  Arms: Non-Accelerated

SUMMARY:
This study is comparing accelerated versus nonaccelerated rehabilitation following ACL reconstruction. Patients undergoing ACL reconstruction will be randomly allocated to one of the two rehabillitation pathways. They will then be monitored over a 15 month period.

DETAILED DESCRIPTION:
The anterior cruciate ligament (ACL) is a vital structure within the knee that provides the stability of the joint. Injury to the ACL is a common injury of the knee affecting young adults, usually whilst playing sport.

Surgical reconstruction of complete ACL rupture aims to restore stability of the knee, reduce pain and swelling, limit future arthritic change, maximise knee function and allow patients to return to preinjury recreational and sporting activity. It has been suggested that the success of an ACL reconstruction is dependent upon the postoperative rehabilitation process.

There is no consensus on the best rehabilitation following ACL reconstruction. Traditional, nonaccelerated, rehabilitation programmes emphasise protection of the ACL graft, modelled on the stages of graft healing. This includes postoperative immobilisation, limiting how much the knee can be straightened, restricted weight bearing and delayed return to activity with most patients returning to activity at 1 year. Complications have however been identified with nonaccelerated rehabilitation. This includes ongoing muscle weakness, inability to fully straighten the knee, and knee cap pain at 1 year followup. To address these issues alternative, accelerated, rehabilitation programmes have been developed. These have included allowing full movement, earlier weight bearing and earlier return to activity, with no adverse sequalae.

The uncertainty in the benefit of accelerated rehabilitation over conventional nonaccelerated protocols warrants further investigation in order determine whether accelerated protocols improve knee muscle function and clinical outcome in the longterm, and provide a more effective practice for treating patients following ACL reconstruction, or whether they pose an increased risk of reinjury by permitting early return to higher level activity.

This study is a single centre randomized controlled trial comparing accelerated versus nonaccelerated rehabilitation protocols with the use of clinical and patient reported outcome measures over a 15month period following ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 16 years or over, listed for primary ACL reconstruction using hamstring grafts at North Bristol NHS Trust.

Exclusion Criteria:

* Patients listed for double bundle ACL reconstruction.
* Patients listed for multiple ligament reconstruction.
* Patients listed for revision reconstructive surgery of the knee.
* Previous history of lower limb arthroplasty.
* Previous history of knee injury in either knee, e.g. meniscal tears, previous ligament injuries.
* Patients unable to understand or read English (the outcome measures being utilised have been validated or published in the English language only).
* Patients unable to comply with the study protocol.
* Patients unable to attend for rehabilitation at North Bristol NHS Trust.
* Meniscal repairs resulting in subsequent modification to the rehabilitation protocol (e.g. altered weight bearing, brace).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09-19 (Actual); Study Completion 2016-09-19 (Actual)

PRIMARY OUTCOMES:
IKDC data completion | 15 months
  As a measure of the feasibility of the study design
KOOS data completion | 15 months
  As a measure of the feasibility of the study design
Tegner data completion | 15 months
  As a measure of the feasibility of the study design
EQ5D data completion | 15 months
  As a measure of the feasibility of the study design
Anterior/Posterior knee translation completion | 15 months
  As a measure of the feasibility of the study design
Lower Limb Symmetry completion | 15 months
  As a measure of the feasibility of the study design

CONTACTS AND LOCATIONS:
Overall Officials: James Robinson, MBBS, FRCS (Orth), Principal Investigator — North Bristol NHS Trust
Locations (1):
- North Bristol NHS Trust, Bristol, United Kingdom